CLINICAL TRIAL: NCT07262892
Title: Three-Dimensional Evaluation of the Effects of Different Maxillary Expansion Methods
Brief Title: 3D Evaluation of Maxillary Expansion Methods
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Büşra Zeynep Yörük (Other)
Collaborators: Centerdent Orthodontics & Aesthetic Dentistry Clinic (Unknown)
Responsible Party: Sponsor-Investigator, Büşra Zeynep Yörük, Phd Student, Bezmialem Vakif University
Organization: Bezmialem Vakif University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E.181356
Record Dates: First submitted 2025-11-21; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Maxillary Transverse Deficiency
Keywords: Maxillary Expansion; Rapid Maxillary Expansion (RME); Invisalign Palatal Expander (IPE); Transverse Maxillary Deficiency; Three-Dimensional Evaluation; Orthodontics; Pediatric Dentistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IPE Group (Experimental): Participants in this group will receive treatment with the Invisalign Palatal Expander (IPE). Three-dimensional (3D) intraoral and extraoral scans will be taken at the end of expansion, at 3 months, and at 6 months.
  Interventions: Device: Invisalign Palatal Expander (IPE)
- RME Group (Experimental): Participants in this group will receive treatment with an acrylic cap splint Rapid Maxillary Expansion (RME) appliance. Three-dimensional (3D) intraoral and extraoral scans will be taken at the end of expansion, at 3 months, and at 6 months.
  Interventions: Device: Acrylic Cap Splint Rapid Maxillary Expansion (RME) Appliance
- Control Group (No Intervention): Participants in this group will not receive orthodontic expansion treatment during the study period and will serve as untreated controls. 3D intraoral and extraoral scans will be obtained at the same time points as treatment groups (end of expansion period equivalent, 3 months, 6 months).

INTERVENTIONS:
Device: Invisalign Palatal Expander (IPE) — A removable, nylon palatal expander produced via digital workflow and 3D printing. Activations are planned at 0.25 mm per activation according to manufacturer protocol. Device is fitted to palatal curvature and used until desired expansion achieved, followed by retention.
  Arms: IPE Group
Device: Acrylic Cap Splint Rapid Maxillary Expansion (RME) Appliance — Bonded acrylic cap splint RME with a jackscrew activated typically at 0.5 mm per day until expansion goal is reached, followed by retention period. Used in pediatric orthodontic practice.
  Arms: RME Group

SUMMARY:
This controlled prospective clinical trial aims to evaluate the effectiveness of different maxillary expansion methods in children with maxillary transverse deficiency. A total of 60 participants will be included: 20 patients will receive Invisalign Palatal Expander (IPE), 20 will receive acrylic cap splint Rapid Maxillary Expansion (RME), and 20 will serve as an untreated control group. Three-dimensional (3D) intraoral and extraoral scans will be taken at the end of expansion, at 3 months, and at 6 months. Primary outcomes include maxillary arch width, first molar angulation, palatal surface area, and palatal volume. Secondary outcomes include soft tissue changes in the facial region. This study provides a direct comparison between a traditional and a modern digital expansion method, generating evidence for clinical decision-making in pediatric orthodontics.

DETAILED DESCRIPTION:
Maxillary transverse deficiency is a common craniofacial problem that often presents with posterior crossbite and dental crowding. Rapid Maxillary Expansion (RME) achieves sutural separation and bone remodeling, typically activated at 0.5 mm per day. Invisalign® Palatal Expander (IPE) is a modern digital system using 3D printing to produce removable nylon expanders adapted to palatal curvature, with 0.25 mm activations, simplifying oral hygiene and eliminating screw activation.

This controlled prospective clinical trial will recruit 60 children with maxillary transverse deficiency. Participants will be assigned to three groups: IPE (n=20), RME (n=20), and untreated control (n=20). Intraoral scans will be obtained at the end of expansion, at 3 months, and at 6 months to create three-dimensional digital models. Maxillary dental arch widths, first molar angulations, palatal surface areas, and volumes will be measured. Extraoral 3D facial scans will evaluate soft tissue changes, including nasal tip, alar width, and interzygomatic distance.

Statistical analyses will be performed using SPSS, applying t-tests for intra- and inter-group comparisons. The study aims to provide comparative data on a traditional (RME) and a contemporary digital (IPE) maxillary expansion method. No prior studies have directly compared these two techniques in children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-12 years
* Good oral hygiene and adequate patient cooperation
* No previous orthodontic expansion treatment

Exclusion Criteria:

* Systemic diseases affecting growth, bone metabolism, or craniofacial development
* Craniofacial syndromes or congenital anomalies
* Severe behavioral or cooperation problems
* Previous orthodontic or orthopedic maxillary expansion
* Patients undergoing medications that affect bone metabolism

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Maxillary First Molar Tipping | Baseline (T0), 3 months after expansion (T1), and 6-month retention period (T2)
  The angulation of the maxillary first molars will be measured using three-dimensional digital models obtained at T0, at 3 months after completion of expansion (T1), and at the 6-month retention follow-up (T2). Angular changes will be calculated through superimposition of maxillary 3D models and standardized angular measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) from this study, including intraoral and extraoral 3D scans, radiographs will be made available to other researchers upon reasonable request. All data will be anonymized to protect patient confidentiality. Access requests will be reviewed by the principal investigator, and researchers will be required to sign a data use agreement to ensure appropriate and secure use of the data.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available beginning 6 months after publication of the study results, for a period of 5 years.
Access Criteria: De-identified individual participant data (IPD), including intraoral and extraoral 3D scans, radiographs along with the study protocol, statistical analysis plan, and analytic code, will be available to qualified researchers. Access will be granted upon reasonable request, reviewed by the principal investigator. Researchers must submit a proposal and sign a data use agreement to ensure confidentiality and appropriate use of the data. Data will be shared through a secure repository after publication of the primary results.
URL: https://bezmialem.edu.tr/en/Pages/academic/clinical/Clinical-Research-Ethics-Committee.aspx

REFERENCES:
- [Result] Bruni A, Ferrillo M, Gallo V, Parrini S, Garino F, Castroflorio T, Deregibus A. Efficacy of clear aligners vs rapid palatal expanders on palatal volume and surface area in mixed dentition patients: A randomized controlled trial. Am J Orthod Dentofacial Orthop. 2024 Sep;166(3):203-214. doi: 10.1016/j.ajodo.2024.04.006. Epub 2024 Jul 26. PMID 39066746
- [Result] Turker G, Coban G, Bayraktar AU, Kurt G, Kilic E, Alkan A. Three-dimensional palatal morphology and upper arch changes following nonsurgical and surgical maxillary expansion in adults. Oral Surg Oral Med Oral Pathol Oral Radiol. 2022 Oct;134(4):425-431. doi: 10.1016/j.oooo.2022.02.013. Epub 2022 Mar 3. PMID 35490136